CLINICAL TRIAL: NCT06962436
Title: Robotic-Assisted Bronchoscopy Versus Ultrathin Bronchoscope Combined With Virtual Bronchoscopic Navigation for the Diagnosis of Peripheral Pulmonary Nodules: A Prospective, Multicenter, Randomized Controlled，Non-inferiority Clinical Study
Brief Title: RAB Versus Ultrathin Bronchoscopy With VBN in the Diagnosis of PPNs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Deputy Hospital Director, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE202503
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAB group (Experimental): The eligible patient will be diagnosed using the robotic bronchoscopy system and catheters developed by Changzhou Langhe Medical Devices Co., Ltd.
  Interventions: Device: Robotic bronchoscopy system
- UB-VBN group (Active Comparator): The eligible patient will be diagnosed using ultrathin bronchoscope combined with virtual bronchoscopic navigation.
  Interventions: Device: Ultrathin bronchoscope combined with virtual bronchoscopic navigation

INTERVENTIONS:
Device: Robotic bronchoscopy system — Utilization of a robotic bronchoscopy system for the biopsy of patients with peripheral pulmonary lesions suspected of malignancy
  Arms: RAB group
Device: Ultrathin bronchoscope combined with virtual bronchoscopic navigation — Utilization of ultrathin bronchoscope combined with virtual bronchoscopic navigation for the biopsy of patients with peripheral pulmonary lesions suspected of malignancy
  Arms: UB-VBN group

SUMMARY:
The purpose of this study is to evaluate whether the diagnostic yield of robotic-assisted bronchoscopy is not inferior to that of the virtual bronchoscopic navigation combined with ultrathin bronchoscopy.

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, multicenter, randomized , non-inferiority clinical trial, with a total of 184 participants planned for enrollment. Subjects with peripheral pulmonary nodules (PPNs) suspected of malignancy, requiring non-surgical biopsy detected by chest CT will be included in this study. Firstly, the physician will determine the lesion to be biopsied, then the subject will be randomly assigned to either the experimental or control group. The experimental group will undergo the procedure using the robotic-assisted bronchoscopy system and catheters, developed by Changzhou Langhe Medical Devices Co., Ltd. for the localization and sampling of PPNs. The control group will undergo ultrathin bronchoscopy guided by virtual bronchoscopic navigation. Radial endobronchial ultrasound (r-EBUS) will be available for all procedures. If the physician determines that biopsy sampling is feasible, a transbronchial lung biopsy will be performed. The primary endpoint is the diagnostic yield. Secondary endpoints include navigation success yield, arrival time, and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of gender;
2. Patients with peripheral lung nodules of suspected malignancy on chest CT who require non-surgical biopsy;
3. Patients who voluntarily consent to undergo bronchoscopy and meet the requirements for the bronchoscopy;
4. Patients should understand the purpose of the trial, demonstrate good compliance with the examinations and follow-ups, and voluntarily participate in the clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Presence of contraindications for bronchoscopy, including: active massive hemoptysis; recent myocardial infarction or unstable angina; severe cardiac or pulmonary dysfunction; severe hypertension and arrhythmias; uncorrectable bleeding tendencies or severe coagulation disorders (such as platelet count <60×10^9/L), uremia; severe pulmonary artery hypertension; severe superior vena cava syndrome; intracranial hypertension; acute cerebrovascular events; aortic dissection or aneurysm; multiple bullae; extreme systemic exhaustion;
2. Patients with pure ground-glass nodules suspected of malignancy on chest CT;
3. Female patients who are breastfeeding, pregnant, or planning pregnancy;
4. Patients with electromagnetic active implantable medical devices;
5. Subjects allergic to anesthetics; or with a history of multiple severe allergies, hereditary allergy history;
6. Those who have participated in or are currently participating in drug clinical trials within 3 months before screening, or have participated in other medical device clinical trials within 30 days;
7. Any other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 14 days post-procedure
  Diagnostic yield= (number of nodules diagnosed with malignancies or specific benign results by study procedure / total number of nodules biopsied by bronchoscopy in each group) * 100%

SECONDARY OUTCOMES:
Navigation success yield | During the procedure
  Navigation success yield = (number of nodules successfully navigated / total number of nodules biopsied by bronchoscopy in each group) * 100%
Navigation time | During the procedure
  In the experimental group, the navigation time is measured from the tracheal carina after the registration to the moment the lesion is visible at the front-end camera of the catheter or confirmed by r-EBUS. In the control group, the navigation time is measured from the tracheal carina to the moment the lesion is confirmed by r-EBUS.
Incidence of complications | 14 days post-procedure
  Incidence of complications = (number of cases with complications / total number of sampled cases) * 100%.
  Complications are categorized according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and include events such as pneumothorax and bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (5):
- China (5):
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital , affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No